CLINICAL TRIAL: NCT06971692
Title: Transdiagnostic Therapy With Metacognitive Therapy Versus Unified Protocol for Patients With Comorbid Anxiety Disorders: a Randomized Controlled Trial
Brief Title: Metacognitive Therapy vs Unified Protocol for Patients With Comorbid Anxiety Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Fredrik Santoft, Lic. psychologist, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-01509-01
Record Dates: First submitted 2025-04-25; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Generalized Anxiety Disorder (GAD); Social Anxiety Disorder (SAD); Panic Disorder (With or Without Agoraphobia)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Generalized Anxiety Disorder; Phobia, Social; Panic Disorder

STUDY DESIGN:
Intervention Model Description: Participants are consecutively recruited and randomly allocated to conditions using a 1:1 ratio.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors conducting diagnostic interviews and clinical severity ratings, at post and follow-up assessments, are blinded to treatment condition and baseline diagnostic status.
  Investigators are blinded to treatment condition in the analysis phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metacognitive therapy (MCT) (Experimental): Transdiagnostic MCT, focused on modifying dysfunctional metacognitions and thereby reducing attentional and cognitive processes central to maintaining anxiety disorders.
  Interventions: Behavioral: Metacognitive therapy (MCT)
- Unified protocol (UP) (Active Comparator): Transdiagnostic cognitive-behavioral therapy, focused on emotion regulation processes central to the development and maintenance of anxiety disorders, particularly neuroticism.
  Interventions: Behavioral: Unified protocol (UP)

INTERVENTIONS:
Behavioral: Metacognitive therapy (MCT) — MCT is delivered in weekly face-to-face sessions
  Arms: Metacognitive therapy (MCT)
Behavioral: Unified protocol (UP) — UP is delivered in weekly face-to-face sessions
  Arms: Unified protocol (UP)

SUMMARY:
The primary goal of this randomized controlled trial is to compare the effectiveness of two transdiagnostic psychological treatments, Metacognitive Therapy (MCT) and the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP), for patients with complex anxiety.

DETAILED DESCRIPTION:
Background:

Anxiety disorders are highly prevalent, impairing quality of life and contributing to substantial economic burden. A large portion of the affected individuals also fulfill the criteria for at least one other anxiety disorder and/or depression. This comorbidity is associated with increased symptom severity and a poorer prognosis. Cognitive-behavioral therapy (CBT) is effective but traditionally relies on a specific manual for every distinct disorder, complicating the management of comorbidity and increasing training needs for therapists. Transdiagnostic therapies target underlying, shared mechanisms across anxiety disorders and depression, and can be used regardless of specific diagnoses. They thereby offer potential for efficient treatment of complex presentations, addressing a wider range of patients' problems with simplified therapist training.

Aims:

The primary aim of the study is to compare the effectiveness of two transdiagnostic therapies, MCT and UP, for patients with comorbid anxiety. Beyond evaluating effectiveness, the project seeks to identify the key factors that drive improvement during treatment. Research questions:

1. Are there differences in effect between MCT and UP regarding clinician-rated severity of anxiety and depression diagnoses after treatment?
2. Are there differences in effect between MCT and UP regarding patients' self-reported symptoms of anxiety, depression, and functioning after treatment?
3. Are there differences in effect between MCT and UP regarding clinician-rated severity of anxiety and depression diagnoses, as well as patients' self-reported symptoms of anxiety, depression, and functioning, at the 1-year follow-up after completed treatment?
4. Does improvement occur in patients in the way that the treatment methods (MCT and UP, respectively) are intended to work, according to the presumptive mechanisms of change?

Methods:

* Design and participants: Patients (N = 114) are randomly allocated in a 1:1 ratio to MCT or UP. Patients are consecutively recruited from the regular influx at two psychiatric clinicis in Stockholm, Sweden. See sections Study design and Eligibility.
* Measurements: Most measures are rated at baseline, post-treatment and at the 1-year follow-up. For the purpose of mediational analyses, procsess measures as well as outcome measures of anxiety and depression are rated weekly during treatment. See section Outcome Measures.
* Treatment conditions: Treatment (MCT or UP) is delivered in approximately 10-18 weekly face-to-face sessions. See section Arms and Interventions.
* Data analyses: Analyses of treatment effects, including the primary outcome of pre- to post changes in Clinical Severity Rating (CSR) between conditions, are conducted according to the intention-to treat principle, using multilevel modeling. Model-based effect sizes, with 95% confidence intervals, are also calculated. For assessment of treatment response, disorder-specific measures are used with criteria for reliable change and clinical cut-off, rendering the categories recovered, improved, unchanged, or deteriorated. Remission status is also assessed according to blinded clinician-rated severity of anxiety and depression diagnoses after treatment, where CSR < 4 means that a patient no longer fulfills criteria for a diagnosis. Differences in proportions are evaluated with chi-squared tests. Mediational analyses are conducted by disaggregating potential mediators to their within- and between-person components. To establish a temporal sequence between mediator and outcome, mediator scores are lagged relative to outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Ability to read and speak Swedish
* A principal diagnosis of post-traumatic stress disorder, generalized anxiety disorder, social anxiety disorder, or panic disorder
* At least one additional comorbid diagnosis (one of the above diagnoses, or obsessive-compulsive disorder, or major depressive disorder)
* Patients on psychotropic medication must have been on a stable dose (excluding as-needed medication) for at least six weeks prior to treatment initiation

Exclusion Criteria:

* Current diagnosis of psychosis, bipolar disorder or moderate to severe substance use disorder
* Medium to high suicide risk
* Psychiatric, somatic or social problems that require primary intervention other than the treatments offered in the study
* Concurrent psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Severity Rating (CSR): change over time | Baseline, post-treatment (immediately after treatment completion of up to 18 weeks/sessions), 1-year follow-up.
  Diagnoses are assigned a dimensional clinical severity rating on a scale from 0 (no symptoms) to 8 (extremely severe symptoms), with a rating of 4 or higher representing the clinical threshold for diagnostic criteria. Observer-assessed.

SECONDARY OUTCOMES:
Overall Anxiety Severity and Impairment Scale (OASIS): change over time | Baseline, weekly during treatment (through up to 18 weeks/sessions) post-treatment (immediately after treatment completion of up to 18 weeks/sessions), 1-year follow-up
  Self-reported anxiety
Overall Depression Severity and Impairment Scale (ODSIS): change over time | Baseline, weekly during treatment (through up to 18 weeks/sessions) post-treatment (immediately after treatment completion of up to 18 weeks/sessions), 1-year follow-up
  Self-reported depression
Generalized Anxiety Disorder-7 (GAD-7): change over time | Baseline, post-treatment (immediately after treatment completion of up to 18 weeks/sessions), 1-year follow-up
  Self-reported anxiety
Patient Health Questionnaire-9 (PHQ-9): change over time | Baseline, post-treatment (immediately after treatment completion of up to 18 weeks/sessions), 1-year follow-up
  Self-reported depression
Posttraumatic Stress Disorder Checklist-5 (PCL-5): change over time | Baseline, post-treatment (immediately after treatment completion of up to 18 weeks/sessions), 1 year follow-up
  Self-reported symptoms of post-traumatic stress. Only for patients with a principal diagnosis of Posttraumatic Stress Disorder.
Penn State Worry Questionnaire (PSWQ): change over time | Baseline, post-treatment (immediately after treatment completion of up to 18 weeks/sessions), 1 year follow-up
  Self-reported symptoms of generalized anxiety. Only for patients with a principal diagnosis of Generalized Anxiety Disorder.
Liebowitz Social Anxiety Scale-Self-Report (LSAS-SR): change over time | Baseline, post-treatment (immediately after treatment completion of up to 18 weeks/sessions), 1 year follow-up
  Self-reported symptoms of social anxiety. Only for patients with a principal diagnosis of Social Anxiety Disorder.
Panic Disorder Severity Scale-Self-Rated (PDSS-SR): change over time | Baseline, post-treatment (immediately after treatment completion of up to 18 weeks/sessions), 1 year follow-up
  Self-reported symptoms of panic. Only for patients with a principal diagnosis of Panic Disorder.
World Health Organization Disability Assessment Schedule (WHODAS-12): change over time | Baseline, post-treatment (immediately after treatment completion of up to 18 weeks/sessions), 1-year follow-up
  Self-reported functional impairment
Difficulties in Emotion Regulation Scale-16 (DERS-16): change over time | Baseline, weekly during treatment (through up to 18 weeks/sessions) post-treatment (immediately after treatment completion of up to 18 weeks/sessions)
  Self-reported difficulties in emotion regulation. Process measure.
Cognitive Attentional Syndrome (CAS-1): change over time | Baseline, weekly during treatment (through up to 18 weeks/sessions) post-treatment (immediately after treatment completion of up to 18 weeks/sessions)
  Self-reported cognitive attentional syndrome and metacognitions. Process measure.
Metacognitions Questionnaire-30 (MCQ-30) - subscale danger and uncontrollability: change over time | Baseline, weekly during treatment (through up to 18 weeks/sessions) post-treatment (immediately after treatment completion of up to 18 weeks/sessions)
  Self-reported metacognitions. Process measure.
Credibility/Expectancy Questionnaire (CEQ): after session 3 | After session 3 (between week 3 and 4)
  Self-reported credibility of treatment and expectancy of improvement
Facilitative Interpersonal Skills scale for Clients (FIS-C): after session 3 | After session 3 (between week 3 and 4)
  Self-reported perspectives on therapist characteristics
Negative Effects Questionnaire (NEQ): after treatment | Post-treatment (immediately after treatment completion of up to 18 weeks/sessions)
  Self-reported adverse events
Client Satisfaction Questionnaire (CSQ): after treatment | Post-treatment (immediately after treatment completion of up to 18 weeks/sessions)
  Self-reported satisfaction with treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Psykiatri Nordväst and Psykiatri Sydväst, Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No